CLINICAL TRIAL: NCT02623920
Title: Phase II Study of Brentuximab Vedotin in Combination With Bendamustine and Rituximab, in Patients With CD30 Positive, Relapsed or Refractory B Cell Non-Hodgkin Lymphoma (NHL)
Brief Title: Brentuximab Vedotin, Bendamustine, and Rituximab in Patients With Relapsed or Refractory B-cell Non-Hodgkin Lymphoma
Acronym: S-BR
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Pharmaceutical company supplying the drug withdraw financial support. PI has decided to close study prior to enrollment of any patients.
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1507953455
Record Dates: First submitted 2015-09-24; First posted 2015-12-08 (Estimated); Last update posted 2017-05-19 (Actual); Status verified 2017-05

CONDITIONS: Diffuse Large B Cell Lymphoma; Mediastinal Large B-cell Lymphoma; Grey Zone Lymphoma; High Grade B Cell Lymphoma; Follicular Lymphoma; Marginal Zone Lymphoma; Small Lymphocytic Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Lymphoma, Follicular; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Brentuximab Vedotin; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Brentuximab, Bendamustine, Rituximab (Experimental): Brentuximab Vedotin in Combination with Bendamustine and Rituximab
  Interventions: Drug: Brentuximab; Drug: Bendamustine; Drug: Rituximab

INTERVENTIONS:
Drug: Brentuximab — Brentuximab vedotin IV over 30 minutes on day 1.Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Other Names: Brentuximab Vedotin; Adcetris
Drug: Bendamustine — Bendamustine IV over 30-60 minutes on days 1-2. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Other Names: Treanda
Drug: Rituximab — Rituximab IV on day 2. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Other Names: Rituxan

SUMMARY:
This phase II trial studies how well brentuximab vedotin, bendamustine, and rituximab work in treating patients with B-cell non-Hodgkin lymphoma that has returned after a period of improvement or has not responded to previous treatment. Monoclonal antibody-drug conjugates, such as brentuximab vedotin, use antibody to target chemotherapy in cancer cells. Drugs used in chemotherapy, such as bendamustine, work in different ways to kill cancer cells. Monoclonal antibodies, such as rituximab, kill the cancer cells directly, but also harness the immune system to kill the cancer cells. Adding brentuximab to rituximab may improve response rates in CD30 positive, CD20 positive Relapsed Refactory NHL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Complete response (CR) rate and overall response rate (ORR) for patients with relapsed aggressive high-risk non-Hodgkin lymphoma (NHL) treated with brentuximab vedotin, bendamustine and rituximab (S-BR).

SECONDARY OBJECTIVES:

I. To estimate 2-year progression-free survival (PFS). II. To evaluate rate of positron emission tomography (PET)-CR and correlation to 2 year PFS.

III. To evaluate the toxicity of six cycles of S-BR. IV. To evaluate mobilization, stem cell collection, engraftment in patients that proceed to salvage autologous stem cell transplant (ASCT).

SCIENTIFIC OBJECTIVES:

I. To evaluate percentage of tumor cells that are positive or negative for cluster of differentiation (CD)30 by immunohistochemistry (IHC), the subcellular location of CD30 (membrane or cytoplasmic only with absence of membrane expression), intensity of scoring, and correlating with clinical outcomes.

II. To evaluate gene expression profiling (GEP) by Nanostring Technology and comparing expression levels of target genes in CD30 membrane positive, CD30 cytoplasmic only positive or CD30 negative tumor cells.

III. To evaluate correlation between mutations identified through next generation sequencing (NGS) including ribonucleic acid (RNA) sequencing of the tumor transcriptome, and correlating to GEP and CD30 IHC, and correlating to clinical outcomes.

IV. To evaluate the levels of soluble CD30 at baseline and in response to treatment.

SCHEDULE:

Patients receive brentuximab vedotin intravenously (IV) over 30 minutes on day 1, bendamustine IV over 30-60 minutes on days 1-2, and rituximab IV on day 2. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* CD30 detectable B lineage relapsed refractory NHL including the following histologies:

  * Aggressive lymphomas: diffuse large B cell lymphoma, primary mediastinal B cell lymphoma, grey zone lymphomas, high grade B cell lymphomas, and transformed indolent lymphomas
  * Indolent lymphoma: follicular lymphoma, marginal zone lymphoma, small lymphocytic lymphoma; indolent lymphoma patients eligible for this trial should have high tumor burden and high risk disease, as defined by:

    * The Groupe d'Etude des Lymphomes Folliculaires (GELF) criteria
    * Intermediate or high risk by Follicular Lymphoma International Prognostic Index (FLIPI) score or elevated lactose dehydrogenase (LDH)/ beta-2 microglobulin (B2M)
* Subjects between 18 and 75 years old. Subjects older than 75 years old to be discussed with PI prior to subject consent; consensus between PI and treating physician is required.
* Karnofsky performance status (KPS) >= 70%, Eastern Cooperative Oncology Group (ECOG) =< 2
* At least 1 measurable site of disease according to Revised Response Criteria for Malignant Lymphoma
* Patients must have received at least one but no more than 4 prior lines of systemic therapy
* American Heart Association (AHA) class 1 without significant limitation of physical activity
* Ejection fraction (EF) of at least >= 40% by multigated acquisition (MUGA) or echocardiography (ECHO)
* Total bilirubin =< 1.5 mg/dl
* Alanine aminotransferase (ALT), aspartate aminotransferase (AST) less than 2.5 times the upper limit of normal without evidence of active infectious hepatitis
* Creatinine clearance >= 40 ml/min
* Platelets > 75,000 cells/ul
* Absolute neutrophil count (ANC) > 1,000 cells/ul
* Ability to provide informed consent
* Females of childbearing potential must have a negative serum or urine beta-human chorionic gonadotropin (HCG) pregnancy test at screening; pregnancy testing is not required for: (a) women who have been post-menopausal for at least 2 years without menses; or (b) women who are surgically sterile (e.g. by means of hysterectomy, tubal ligation, etc.)
* Males and females of childbearing potential must be able and willing to use an effective contraceptive method during treatment and for three months after completing treatment

Exclusion Criteria:

* Active infections (bacterial, fungal, or viral)
* Evidence of sanctuary site involvement by disease, e.g., central nervous system, ocular, testicular involvement
* Evidence of second malignancy, abnormal cytogenetics, or morphologic evidence of myelodysplastic syndromes (MDS)
* Recent chemotherapy within 3 weeks of screening
* Major surgery within 4 weeks of screening
* Diagnosed or treated for malignancy other than NHL for which patient will be treated, except: malignancy treated with curative intent and with no known active disease present for >= 3 years before subject registration; adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease; adequately treated carcinoma in situ without evidence of disease
* History of stroke or intracranial hemorrhage within 6 months prior to registration
* Requires anticoagulation with warfarin or equivalent vitamin K antagonists
* Requires treatment with strong cytochrome (CYP3A4/5) inhibitors
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of screening, or any class 3 (moderate) or class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification
* Known history of human immunodeficiency virus or active hepatitis C virus or active hepatitis B virus infection or any uncontrolled active systemic infection requiring intravenous antibiotics
* Women who are pregnant or breastfeeding
* Prior use of brentuximab vedotin
* Prior use of bendamustine for indolent lymphoma allowed if > 2 years, CR to bendamustine and well tolerated with no residual > grade 1 toxicity; no prior use of bendamustine for aggressive lymphoma allowed
* Prior allogeneic transplant
* Patients with Child-Pugh B or C hepatic impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12-16 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
CR rate | Up to 2 years after completion of study treatment
  The complete response rate will be estimated as the proportion of patients with response, with a 95% exact confidence interval.
Percentage of patients obtaining a CR + PR using Cheson criteria | Up to 2 years after completion of study treatment
  The overall response rate will be estimated as the proportion of patients with response, with a 95% exact confidence interval.

SECONDARY OUTCOMES:
Median time to progression | At 2 years
PFS | At 2 years
  PFS will be estimated using the Kaplan-Meier estimate, with stratification by allogeneic stem cell transplantation status.
Complete response rate assessed by PET/CT | Up to 2 years after the completion of study treatment
  The complete response rate by PET/CT will be estimated with the 95% exact confidence interval.
Frequency of adverse events (AEs) and serious AEs assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 2 years after completion of study treatment
  The proportion of patients with treatment-emergent AEs will be tabulated, including by causality, seriousness, severity/grade, and whether the AE resulted in death or discontinuation of treatment.
CD34+ peripheral blood stem cells assessed by flow cytometry | Up to 2 years after completion of study treatment
  Only for subjects receiving transplant
Median time to engraftment | Up to 2 years after completion of study treatment
  Only for subjects receiving transplant
Soluble CD30 levels in blood by biochemical assay | 48-72 hours after brentuximab vedotin treatment
  Brentuximab vedotin pharmacokinetics in combination therapy will be measured and correlated to single agent data.

OTHER OUTCOMES:
CD30 expression by immunohistochemistry (IHC) | Up to 2 years after completion of study treatment
  Subcellular location or CD30 (membrane or cytoplasmic only), intensity of scoring, and association with progression-free survival will be evaluated. These relationships will be assessed using a Cox proportional hazards model. Expression levels of target genes based on CD30 location will be assessed using two sample independent t tests, with adjustment for multiple comparisons to protect the false discovery rate.
Genetic mutations identified by NGS | Up to 2 years after completion of study treatment
  The relationship between mutations identified through next generation sequencing, gene expression profiling, CD30 IHC and progression-free survival will be assessed using a Cox proportional hazards models.
GEP by Nanostring Technology | Up to 2 years after completion of study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Daniel O. Persky, MD, Principal Investigator — University of Arizona
Locations (1):
- Arizona Cancer Center at UMC North, Tucson, Arizona, United States